CLINICAL TRIAL: NCT00005639
Title: A Phase I Dose Escalation to Maximally Tolerated Dose Trial of 5-Azacytidine (5 AC, NSC 102816) in Combination With Sodium Phenylbutyrate (PB, NSC 657802) in Patients With Refractory Solid Tumors
Brief Title: Azacitidine Plus Phenylbutyrate in Treating Patients With Advanced or Metastatic Solid Tumors That Have Not Responded to Previous Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J9982; U01CA070095 (NIH); R01CA075525 (NIH); P50CA058236 (NIH); P30CA006973 (NIH); CDR0000067799; NCI-270; 99-12-03-02 (Other: JHM IRB)
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; unspecified adult solid tumor, protocol specific; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; intraocular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Azacitidine; 4-phenylbutyric acid

ARMS (3):
- Regimen A: 14-day 5-AC with intermittent phenylbutyrate (Experimental): Participants receive low-dose regimen of 5-AC with intermittent phenylbutyrate 400 mg/m2/day by continuous intravenous (CIV) over 24 hours on Days 6 and 13. Each cycle lasts 35 days.
  Cohort A1: 25 mg/m2/day subcutaneous (SC) Cohort A-1: 18.75 mg/m2/day SC Cohort A-2: 15 mg/m2/day SC Cohort A-3: 10 mg/m2/day SC
  Interventions: Drug: Azacitidine Injection; Drug: sodium phenylbutyrate
- Regimen B: 7-day 5-AC with sequential phenylbutyrate (Experimental): Participants receive 5-AC 75mg/m2/day SC for 7 days, followed sequentially by two different doses of phenylbutyrate CIV starting on Day 8 and continuing for 7 days. Each cycle lasts 35 days
  Cohort B1: Phenylbutyrate 200 mg/m2/day CIV Cohort B2: Phenylbutyrate 400 mg/m2/day CIV
  Interventions: Drug: Azacitidine Injection; Drug: sodium phenylbutyrate
- Regimen C: 21-day 5-AC with weekly phenylbutyrate (Experimental): Participants receive two different daily doses of 5-AC SC for 21 days and phenylbutyrate 400 mg/m2/day CIV over 24 hours once-per-week. Each cycle lasts 42 days.
  Cohort C1: 5-AC 10mg/m2/day SC Cohort C2: 5-AC 12.5mg/m2/day SC
  Interventions: Drug: Azacitidine Injection; Drug: sodium phenylbutyrate

INTERVENTIONS:
Drug: Azacitidine Injection — subcutaneous injection (SC)
  Other Names: AC; 5-AC
Drug: sodium phenylbutyrate — continuous intravenous (CIV)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of azacitidine plus phenylbutyrate in treating patients with advanced or metastatic solid tumors that have not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the safety and toxicity of azacitidine plus phenylbutyrate in patients with refractory solid tumors.
* Determine the maximum tolerated dose of this treatment regimen where maximal gene reexpression occurs in these patients.
* Evaluate the pharmacokinetics of these drugs in these patients.
* Determine the minimally effective dose of azacitidine in combination with phenylbutyrate that elicits a biological or clinical response in these patients.

OUTLINE: This is a dose escalation study.

Patients receive azacitidine subcutaneously for 14-21 days and sodium phenylbutyrate IV continuously for 1-7 days. Treatment repeats every 35 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses and durations of treatment with azacitidine and phenylbutyrate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities.

PROJECTED ACCRUAL: Approximately 3-50 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
Inclusion criteria:

DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced or metastatic malignant solid tumor not amenable to curative therapy

  * Lymphoma allowed
* Progressive disease
* Evaluable disease
* No CNS metastases by CT scan or MRI

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 8 g/dL (may be achieved by transfusion)
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 mg/dL (unless due to hemolysis or Gilbert's syndrome)
* SGOT and SGPT less than 2 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* No active infection
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 2 weeks before, during, and 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior adjuvant chemotherapy for advanced or metastatic disease and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2000-03 (Actual); Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Minimal Effective Dose (MED) of Azacitidine with Phenylbutyrate | up to 6 months
  MED (milligrams) of combined Azacitidine and Phenylbutyrate that results in clinical response, as defined by Standard World Health Organization (WHO) criteria and/or target inhibition.

SECONDARY OUTCOMES:
Toxicity as assessed by number of participants experiencing adverse events Grade 3 or higher as defined by CTCAE v2.0 | up to 6 months
Pharmacokinetics of Azacitidine combined with Phenylbutyrate as measured by maximal plasma concentration (Cmax) | Up to 24 hours
Gene-re-expression of epigenetic modulation in Peripheral Blood Mononuclear Cells (PBMC) as measured by change in Epstein-Barr Virus (EBV) viral load (number of copies per 1 million cells) after treatment with Azacitidine | Change from baseline to up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Carducci, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Lin J, Gilbert J, Rudek MA, Zwiebel JA, Gore S, Jiemjit A, Zhao M, Baker SD, Ambinder RF, Herman JG, Donehower RC, Carducci MA. A phase I dose-finding study of 5-azacytidine in combination with sodium phenylbutyrate in patients with refractory solid tumors. Clin Cancer Res. 2009 Oct 1;15(19):6241-9. doi: 10.1158/1078-0432.CCR-09-0567. Epub 2009 Sep 29. PMID 19789320